CLINICAL TRIAL: NCT05743426
Title: Disease Outcomes and Toxicities in Patients With Gastrointestinal and Sarcomatous Malignancies
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2247
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Sarcoma; Gastrointestinal Cancer
Keywords: toxicity; survey
MeSH Terms: conditions — Sarcoma; Gastrointestinal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Subjects who are with gastrointestinal malignancies or sarcoma receive radiotherapy.
  Interventions: Other: Survey; Other: Toxicity Assessments

INTERVENTIONS:
Other: Survey — Patient Reported Outcome (PRO) questionnaire
Other: Toxicity Assessments — Toxicity Assessments will be performed using the National Cancer Institute Common Terminology Criteria (NCI-CTCAE).

SUMMARY:
This prospective, single-institution, observational study explores disease outcomes and toxicities in subjects with gastrointestinal malignancies and sarcoma (bone and soft tissue) who are being treated with standard-of-care therapies including radiotherapy.

Recent advances in treatment approaches affected disease outcomes and toxicities. Prospective monitoring of disease outcomes and toxicities using standardized assessments will provide information about recent changes in the standard of care and further refine treatment approaches and prospective clinical trial design.

ELIGIBILITY:
Inclusion Criteria

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Subject is willing and able to provide written informed consent to participate in the study and HIPAA authorization for the release of personal health information. Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designer.
2. Age ≥ 18 years at the time of consent.
3. Histological, cytological, or radiographic evidence/confirmation of a gastrointestinal malignancy or sarcoma.
4. Females with childbearing potential and male subjects with fathering potential are allowed to participate in this study.

Exclusion Criteria

All subjects meeting any exclusion criteria at baseline will be excluded from study participation.

1. Inability or unwillingness to provide informed consent
2. Patients who state they do not expect to be available or willing to follow up at expected intervals post-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with gastrointestinal malignancy or sarcoma receiving treatment at study center.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2036-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Up to 10 years
  Disease-free survival is defined as the length of time after treatment in which the subject survives with no signs or symptoms of cancer.

SECONDARY OUTCOMES:
Local Control | Up to 10 years
  Local Control is defined as radiographic and clinical assessments determined by the patient's treating physician.
Adverse Events | Up to 10 years
  The NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5 is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Quality of life PRO-CTCAE | Up to 10 years
  Quality of life PRO-CTCAE will be evaluated using patient-reported quality of life The PRO-CTCAE is a measurement system that characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities that include pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient's perspective.
  PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present).
Quality of life EQ-5D-5L | Up to 10 years
  Quality of life EQ-5D-5L will be evaluated using EQ-5D-5L. The EQ-5D-5L is a QoL assessment that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels ranging from no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5) to extreme problems.
Quality of life Toronto Extremity Salvage Score (TESS) | Up to 10 years
  Toronto Extremity Salvage Score (TESS) quality of life questionnaire will be used in subjects with sarcoma.
  The TESS is a 30-item patient-reported outcome questionnaire that addresses daily activity limitations including restrictions in body movement, mobility, self-care, and performance of daily tasks. It is scored from 0 (not possible) to 5 (without any problem). Higher scores indicate less functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore K Yanagihara, Principal Investigator — Lineberger Comprehensive Cancer Center, The University of North Carolina Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials